CLINICAL TRIAL: NCT01809730
Title: Pilot Study: Cardiovascular Events in High Risk Orthopedic Surgical Patients
Status: Withdrawn | Type: Observational
Why Stopped: no participants enrolled
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S12-02513
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease; Cerebral Vascular Disease; Peripheral Artery Disease; Renal Insufficiency; Diabetes; COPD; Hypertension; Active Smoker; Cancer; CHF; Prior DVT/PE
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Renal Insufficiency; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Hypertension; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CV biomarkers - inflammatory, metabolic, hypercoagulable and platelet.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiovascular risk: patients with CV disease

SUMMARY:
This is a non-randomized, non-interventional pilot observational study designed to follow high-risk patients through their surgical and hospital stay. The investigators will collect 2 4ml vial's of blood (total of 8ml) prior to surgery to assess CV biomarkers - inflammatory, metabolic, hypercoagulable and platelet.

DETAILED DESCRIPTION:
This study is primarily an observational pilot study. After identifying patients as high-risk according to the following criteria: CAD and/or CVD and/or PAD and/or >=60 years old and at least 2 of the following - renal insufficiency, diabetes, COPD, hypertension, active smoker (or active within 6 months of consent), cancer, congestive heart failure, or any blood clot - they will be asked to sign a consent form. Patients surgical and hospital course will continue as per standard of care. Prior to surgery, 8ml of blood will be collected for to assess cardiovascular biomarkers including inflammatory, metabolic, hypercoagulable and platelet biomarkers to be tested independently in Dr. Berger's lab in Smilow. Study staff will perform electrocardiograms on POD 2. Results of these ECGs will not be placed in the patients' charts. No other procedures will be done for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* • ≥ 21 years of age

  * Subjects undergoing open orthopedic surgery of the hip, knee or spine
  * High-risk subject cohort:
  * Coronary artery disease (CAD), or
  * Cerebrovascular disease (CVD) (prior stroke, TIA or carotid artery disease (>70% stenosis), or
  * Peripheral artery disease (PAD), or
  * Age ≥ 60 years and any 2 of the following:

    * Renal insufficiency (creatinine clearance < 60ml/min)
    * Diabetes
    * Chronic Obstructive Pulmonary Disease (COPD)
    * Hypertension
    * Active smoker or stopped less than 30 days prior to consent
    * Cancer
    * Congestive heart failure
    * Prior blood clot

Exclusion Criteria:

* • Severe co-morbid condition with life expectancy < 6 months

  * Inability to give informed consent or adhere to follow-up as per protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This pilot, observational study is designed to identify and follow orthopedic surgical patients meeting specific high-risk criteria for postoperative cardiovascular events. All normal standard of care will be maintained. Patients will be observed from Pre-Admission Testing (PAT) visit through hospital discharge.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac ischemia/necrosis | 30 days
Venous thromboembolism | 30 days
Pulmonary embolism | 30 dyas
Myocardial infarction | 30 Days
Cerebral vascular event | 30 days
Death | 30 days
Transient ischemic attack | 30 days
Surgical site infection | 30 days
Delayed wound healing | 30 days
Clinically relevant bleeding | 30 days
Transfusion within 48 hours post-op | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Hospital for Joint Diseases, New York, New York, United States